CLINICAL TRIAL: NCT00439881
Title: A Study to Assess the Safety and Tolerability of SB-681323 Administered Via the Intravenous Route
Brief Title: A Study To Look At The Safety Of SB-681323 In Healthy Adult Subjects After Intravenous Administration Of A Single Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RA1107570
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Arthritis, Rheumatoid; Inflammation
Keywords: inflammation,; intravenous,; Chronic Obstructive Pulmonary Disease,; P38 inhibitor; SB-681323,; rheumatoid arthritis,
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation; Pulmonary Disease, Chronic Obstructive | interventions — dilmapimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SB-681323

SUMMARY:
SB-681323 inhibits the action of an enzyme which is known to contribute to the inflammation seen in such conditions as Chronic Obstructive Pulmonary Disease and Rheumatoid Arthritis. This study will explore the safety of this drug and its blood levels when given in intravenous form to healthy human volunteers.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male aged between 25 and 55 years, inclusive, at the time of screening.
* Body weight = 60 kg and a Body Mass Index within the range of 19 to 32 kg/m2 inclusive.
* Must have given informed consent and signed the study consent form prior to taking part in any study procedures.
* Have no significant abnormality on clinical examination.
* Show no abnormality on haematology, clinical chemistry or urinalysis examination at the pre-study medical examination.
* Demonstrate a clinically normal 12-lead ECG at screening
* Liver function tests within the reference range at screening (ALT, AST, ALP, GT and bilirubin)
* Do not show evidence of pre-study HIV and hepatitis B and C at screening
* Do not show a positive pre-study urine drug screen

Exclusion Criteria:

* Taken prescription or over-the-counter medication within 5 days (or 5 half lives, whichever is longer) before the first dosing day, unless the investigator confirms that it will not introduce additional risk or interfere with the study procedures or outcome.
* Show a history or evidence of drug or alcohol abuse.
* Show a history of increased liver function tests (ALT, AST, bilirubin) above upper limit of normal (ULN) in the past 6 months (if known).
* Demonstrate a history of regular alcohol consumption exceeding an average weekly intake of > 21 units (or an average daily intake of greater than 3 units). 1 unit is equivalent to a half-pint (284mL) of beer/lager; 25mL measure of spirits or 125mL of wine.
* Have a history or presence of any medically significant disease, or any disorder that would introduce additional risk or interfere with the study procedures or outcome. In particular, gastro-intestinal, hepatic or renal disease or other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Exposure prior to the first dosing day to more than 3 new medicinal entities within 12 months or has participated in a study with a new medicinal entity within 3 months or any other study within 2 months.
* If participation in the study will result in the subject having donated more than 450 mL blood within a 3 month period.
* On physical examination the subject is observed to have poor venous access.
* An unwillingness of subjects to abstain from sexual intercourse with women; or unwillingness of the subject to use a condom/spermicide in addition to having their female partner use another form of contraception if the woman could become pregnant from the time of the first dose of investigational product until completion of the follow-up procedures.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2006-10

PRIMARY OUTCOMES:
Safety of SB-681323 in terms of frequency/ nature of adverse events and changes in ECG patterns, vital signs and clinical laboratory parameters (including liver function tests) seen upto 48h after a single intravenous dose.

SECONDARY OUTCOMES:
Regular measurements of SB-681323 blood levels upto 48h after a single intravenous dose. Effects of SB-681323 in blood samples drawn upto 24h after intravenous dosing, on laboratory tests designed to explore the anti-inflammatory properties of the drug.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom